CLINICAL TRIAL: NCT04782817
Title: Reducing Reintubation Risk in High-Risk Cardiac Surgery Patients With High-Flow Nasal Cannula
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Freundlich, Assistant Professor of Anesthesiology and Biomedical Informatics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181117
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Intubation; Cardiovascular Surgical Procedure
Keywords: High-flow nasal cannula oxygen therapy; Reintubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Canula Oxygen Therapy (Experimental): Participants will be assigned post extubation physician order set which recommends the administration of oxygen therapy via HFNC. HFNC is a heated and humidified system that allows prescribed fraction of inspired oxygen (FIO2) levels to be delivered at very high flow rates.
  Interventions: Other: Recommendation for high flow nasal cannula oxygen therapy order set
- Provider Choice Standard Care (Active Comparator): Participants be assigned standard provider choice of standard care therapy physician order set.
  Interventions: Other: Provider choice standard care order set

INTERVENTIONS:
Other: Recommendation for high flow nasal cannula oxygen therapy order set — Participants will be assigned post extubation physician order set which recommends the administration of oxygen therapy via HFNC. HFNC is a heated and humidified system that allows prescribed fraction of inspired oxygen (FIO2) levels to be delivered at very high flow rates.
  Arms: High Flow Nasal Canula Oxygen Therapy
Other: Provider choice standard care order set — Participants will receive order set with provider choice of standard care therapy.
  Arms: Provider Choice Standard Care

SUMMARY:
The iCAN trial is a pragmatic randomized controlled trial that aims to test the hypothesis that HFNC versus usual care oxygenation strategies applied immediately after initial extubation after cardiac surgery decreases the all-cause 48-hour reintubation rate (extubation failure within 48 hours of initial extubation).

DETAILED DESCRIPTION:
HFNC may be employed as a strategy to facilitate early extubation and prevent reintubation of patients following cardiac surgery. HFNC is routinely employed by providers in the cardiovascular intensive care unit along with other therapies, including: bi-level positive airway pressure, non-rebreather masks, among others. Currently, no high-quality clinical data exist to demonstrate that HFNC may decrease the risk of reintubation in this critically-ill adult population.

This prospective, randomized, pragmatic clinical trial will compare HFNC to provider choice of usual care in these high-risk patients.

Randomization will occur at the time that the patient is deemed ready for extubation by the attending physician in the cardiovascular intensive care unit. Through randomization, patients will be assigned one of two physician order sets in the electronic medical record system: standard order set with or without recommendation for the use of HFNC. Reintubation and outcome data will be collected until patient discharge.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years
* Undergoing cardiac surgery, defined as a documented surgical service of "cardiac surgery" in the electronic health record, performed in the main operating rooms at Vanderbilt University Medical Center
* Admitted to the cardiovascular intensive care unit postoperatively with an endotracheal tube in place and mechanically ventilated
* Surgery duration (documented time between "Anesthesia start" and "Anesthesia stop" in the EHR) of at least 180 minutes
* Received an order to be extubated by a treating provider o Patients who meet all other criteria but do not receive an order to extubate will be randomized but not enrolled

Exclusion Criteria

• Patient does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reintubation within 48 hours of extubation | 48 hours
  Reintubation within 48 hours of initial extubation after cardiac surgery

SECONDARY OUTCOMES:
Reintubation within 72 hours of extubation | 72 hours
  Reintubation within 72 hours of initial extubation after cardiac surgery
Reintubation after cardiac surgery | hospital discharge (usually 14 days)
  Reintubation at any time during hospitalization after cardiac surgery
All cause mortality | 30 days post surgery
Hospital length of stay | 8 days
Intensive Care Unit length of stay | 3 days
  Intensive Care Unit length of stay after cardiac surgery
Ventilator-free days | 1 day
  Ventilator-free days during hospitalization after cardiac surgery
In-hospital mortality | Until hospital discharge, which usually occurs in approximately 8 days in the majority of patients
  Mortality which occurs in-hospital following surgery, up to the time of hospital discharge
Adjusted reintubation rate | 48 hours
  Adjusted reintubation rate within 48 hours of initial extubation, if adjustment is needed based on clinically relevant imbalance in baseline characteristics between groups

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Freundlich, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khandelwal N, Dale CR, Benkeser DC, Joffe AM, Yanez ND 3rd, Treggiari MM. Variation in tracheal reintubations among patients undergoing cardiac surgery across Washington state hospitals. J Cardiothorac Vasc Anesth. 2015;29(3):551-9. doi: 10.1053/j.jvca.2014.11.009. Epub 2014 Nov 11. PMID 25802193
- [Background] Freundlich RE, Maile MD, Hajjar MM, Habib JR, Jewell ES, Schwann T, Habib RH, Engoren M. Years of Life Lost After Complications of Coronary Artery Bypass Operations. Ann Thorac Surg. 2017 Jun;103(6):1893-1899. doi: 10.1016/j.athoracsur.2016.09.048. Epub 2016 Dec 6. PMID 27938887
- [Background] Dorsa AG, Rossi AI, Thierer J, Lupianez B, Vrancic JM, Vaccarino GN, Piccinini F, Raich H, Bonazzi SV, Benzadon M, Navia DO. Immediate extubation after off-pump coronary artery bypass graft surgery in 1,196 consecutive patients: feasibility, safety and predictors of when not to attempt it. J Cardiothorac Vasc Anesth. 2011 Jun;25(3):431-6. doi: 10.1053/j.jvca.2010.08.013. Epub 2010 Oct 29. PMID 21036063
- [Background] Chan JL, Miller JG, Murphy M, Greenberg A, Iraola M, Horvath KA. A Multidisciplinary Protocol-Driven Approach to Improve Extubation Times After Cardiac Surgery. Ann Thorac Surg. 2018 Jun;105(6):1684-1690. doi: 10.1016/j.athoracsur.2018.02.008. Epub 2018 Mar 9. PMID 29530778
- [Background] Roca O, Hernandez G, Diaz-Lobato S, Carratala JM, Gutierrez RM, Masclans JR; Spanish Multidisciplinary Group of High Flow Supportive Therapy in Adults (HiSpaFlow). Current evidence for the effectiveness of heated and humidified high flow nasal cannula supportive therapy in adult patients with respiratory failure. Crit Care. 2016 Apr 28;20(1):109. doi: 10.1186/s13054-016-1263-z. PMID 27121707
- [Background] Markovitz GH, Colthurst J, Storer TW, Cooper CB. Effective inspired oxygen concentration measured via transtracheal and oral gas analysis. Respir Care. 2010 Apr;55(4):453-9. PMID 20406513
- [Background] Bazuaye EA, Stone TN, Corris PA, Gibson GJ. Variability of inspired oxygen concentration with nasal cannulas. Thorax. 1992 Aug;47(8):609-11. doi: 10.1136/thx.47.8.609. PMID 1412117
- [Background] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Background] Masip J, Peacock WF, Price S, Cullen L, Martin-Sanchez FJ, Seferovic P, Maisel AS, Miro O, Filippatos G, Vrints C, Christ M, Cowie M, Platz E, McMurray J, DiSomma S, Zeymer U, Bueno H, Gale CP, Lettino M, Tavares M, Ruschitzka F, Mebazaa A, Harjola VP, Mueller C; Acute Heart Failure Study Group of the Acute Cardiovascular Care Association and the Committee on Acute Heart Failure of the Heart Failure Association of the European Society of Cardiology. Indications and practical approach to non-invasive ventilation in acute heart failure. Eur Heart J. 2018 Jan 1;39(1):17-25. doi: 10.1093/eurheartj/ehx580. PMID 29186485
- [Background] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Background] Zhu Y, Yin H, Zhang R, Wei J. High-flow nasal cannula oxygen therapy vs conventional oxygen therapy in cardiac surgical patients: A meta-analysis. J Crit Care. 2017 Apr;38:123-128. doi: 10.1016/j.jcrc.2016.10.027. Epub 2016 Nov 9. PMID 27886577
- [Derived] Freundlich RE, Wanderer JP, French B, Moore RP, Hernandez A, Shah AS, Byrne DW, Pandharipande PP. Protocol for a randomised controlled trial: reducing reintubation among high-risk cardiac surgery patients with high-flow nasal cannula (I-CAN). BMJ Open. 2022 Nov 25;12(11):e066007. doi: 10.1136/bmjopen-2022-066007. PMID 36428016